CLINICAL TRIAL: NCT02987413
Title: Safety and Efficacy of Mesenchymal Stem Cells Escalated Application in Amyotrophic Lateral Sclerosis Patients: Study Design of a Phase I Trial
Brief Title: Escalated Application of Mesenchymal Stem Cells in Amyotrophic Lateral Sclerosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital e Maternidade Dr. Christóvão da Gama (Other)
Collaborators: IEP São Lucas - Instituto de Ensino e Pesquisa (Other); Clinica Jordy Sinapse (Unknown); TECHLIFE - Centro de Tecnologia Celular (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HospitalMCG; IEPSaoLucas (Other: IEP Sao Lucas)
Record Dates: First submitted 2016-07-01; First posted 2016-12-09 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Mesenchymal stem cells (Experimental): Two escalated intrathecal infusions of autologous mesenchymal stem cell
  Interventions: Biological: Autologous Mesenchymal stem cells (MSCs)

INTERVENTIONS:
Biological: Autologous Mesenchymal stem cells (MSCs) — 2 intrathecal autologous MSCs infusions (1x10^8 cells) will be performed, escalated from 30 days apart

SUMMARY:
Background: Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease that selectively affects motor neurons in the brain and spinal cord, leading to bulbar, respiratory, and limb weakness. There is no effective treatment, and the disease usually progresses to death within 2 to 4 years. The therapeutic plasticity of mesenchymal stem cells (MSCs) may be an attractive therapy to this complex disease, turning MSCs strong candidates for cellular therapy in ALS.

Design-A phase 1 open-safety clinical trial. 4 patients will be selected according to a restricted inclusion and exclusion criteria and after 2 escalated infusions of MSCs, there will be a follow up period of one year Methods - Primary endpoint: safety of mesenchymal autologous stem cells infusions escalated in two intrathecal administrations in patients with ALS defined as severe adverse events (SAe). Secondary endpoints: clinical response, laboratorial and magnetic resonance imaging of patients submitted to cellular escalating doses applied in the study. Quality of life, according to El Escorial criteria, ALSFR scale and functional scales.

Conclusion: This study is a primary step before a large randomized double-blind clinical trial for ALS. It is expected to confirm the safety of escalated MSCs therapy in ALS patients, initial data of efficacy in addition to improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women and males over 18-year-old.
* Diagnosis of ALS in agreement with the criteria of "EL SCORE"
* Less than 24 months of evolution of the disease (from the beginning of the symptoms).
* Good understanding of the protocol and aptitude to grant the informed consent
* Infertile women (post-menopause or hysterectomized)
* Brazilian citizen and permanent resident.

Exclusion Criteria:

* Any significant medical condition (congestive heart failure, angina, respiratory failure, and others)
* Any auto-immune disease
* Any malignant diseases
* Systemic infection
* Mental illness
* Depressive state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events related to the treatment | 12 months
  Serious Adverse Events (Death, Life-threatening, Disability or Permanent Damage) will be monitored and documented during follow up

SECONDARY OUTCOMES:
Revised ALS Functional Rating Scale (ALSFRS-R) | 12 months
  Quality of life from patients according to functional scales will be evaluated before and after interventions with 1, 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro B Agati, PhD, Study Director — Hospital e Maternidade Dr Christovao da Gama; Eliseo J Sekiya, MD, PhD, Study Chair — Instituto de Ensino e Pesquisas - IEP-São Lucas; Adelson A Silva, MD, Study Chair — Instituto de Ensino e Pesquisas - IEP-São Lucas; Andresa Forte, MSc, Study Chair — TECHLIFE - Centro de Tecnologia Celular; Sergio S Jordy, MD, Study Chair — Clínica Jordy Sinapse
Locations (2):
- Brazil (2):
  - Hospital e Maternidade Dr Christovao da Gama, Santo André, São Paulo
  - Instituto de Ensino e Pesquisas - IEP-São Lucas, São Paulo, São Paulo

REFERENCES:
- See also: Institutional website — http://www.hmcg.com.br